CLINICAL TRIAL: NCT06687408
Title: Sleeve Lobectomy for Lung Cancer in Minimally Invasive Surgical Techniques: a Multicenter Cohort Study
Brief Title: Sleeve Lobectomy for Lung Cancer in Minimally Invasive Surgical Techniques
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Shanghai Chest Hospital of Shanghai Jiao Tong University (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-0959
Record Dates: First submitted 2024-11-08; First posted 2024-11-13 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: lung cancer; sleeve lobectomy; minimally invasive thoracic surgery; perioperative outcomes; long-term survival; robotic-assisted thoracic surgery
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Lung cancer cohort of sleeve lobectomy in minimally invasive surgical approaches: This lung cancer cohort will retrospectively identify and enroll the participants with centrally located primary NSCLC receiving bronchial sleeve resection with or without pulmonary artery angioplasty in minimally invasive approaches (RATS or VATS) between January 2015 and September 2024 from the institutional databases. The choice of minimally invasive surgical approaches depends on the willingness of the surgeons and the participants in this study.
  Interventions: Procedure: RATS Group; Procedure: VATS group

INTERVENTIONS:
Procedure: RATS Group — The participants with centrally located lung cancer in this group were performed sleeve lobectomy in robotic-assisted thoracic surgery (RATS) approach, which has been already applied to these patients in minimally invasive surgical techniques as part of their regular medical care recently.
Procedure: VATS group — The participants with centrally located lung cancer in this group were performed sleeve lobectomy in video-assisted thoracic surgery (VATS) approach.

SUMMARY:
The goal of this multicenter observational study is to evaluate the long-term survival and perioperative outcomes of sleeve lobectomy in robotic-assisted thoracic surgery (RATS) for patients with central lung cancer when compared with video-assisted thoracic surgery (VATS) approach, both of which have been already applied to these patients in minimally invasive surgical techniques as part of their regular medical care recently. The main question it aims to answer is:

Are RATS sleeve lobectomy associated with similar or even better long-term survival and perioperative outcomes for patients with central lung cancer when compared with the VATS approach?

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related deaths worldwide. Approximately 85% of lung cancer is non-small-cell lung cancer (NSCLC). Nowadays, radical surgery resection remains the recommended local treatment for resectable NSCLC, and bronchial and/or pulmonary artery sleeve lobectomy have been proven to be preferred surgical approaches for patients with centrally located lung cancer when compared with traditional pneumonectomy. The long-term survival and perioperative outcomes of sleeve lobectomy in robotic-assisted thoracic surgery (RATS) and video-assisted thoracic surgery (VATS) for central lung cancer were found to be comparable in a few retrospective studies with a limited number of participants. Still, they have not been investigated in the high-volume cohort setting.

Thus, the investigators conducted the multicenter observational cohort study to investigate if RATS sleeve lobectomy was non-inferior to VATS in patients with centrally located NSCLC and to evaluate the long-term survival and perioperative outcomes of sleeve lobectomy in these two regular minimally invasive surgical techniques.

Participants with centrally located primary NSCLC receiving bronchial sleeve resection with or without pulmonary artery angioplasty in minimally invasive approaches (RATS or VATS) between January 2015 and September 2024 were retrospectively identified and enrolled from the institutional database.

In this study, the investigators will focus on the 3-year overall survival (OS) and recurrence-free survival (RFS) of the patients between the two groups (RATS vs. VATS) for the comparison of the long-term oncologic outcomes in the propensity score matching method. Meanwhile, the perioperative outcomes will be investigated between RATS versus VATS sleeve lobectomy, including but not limited to intraoperative blood loss, operative time, length of hospital stay, postoperative drainage, postoperative complications, perioperative mortality, number of dissected lymph nodes, and margin status. In addition, this study will also try to explore the learning curve for RATS sleeve lobectomy and assess the safety and feasibility of minimally invasive sleeve lobectomy in specific patient populations, such as NSCLC patients following neoadjuvant therapy or those with clinical mediastinal lymph node metastasis. Furthermore, the study is designed to summarize the key surgical techniques and practice skills in minimally invasive thoracic surgery to promote technical improvements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Clinically suspected lung cancer with a high likelihood of undergoing sleeve lobectomy;
* Postoperative histopathological diagnosis confirms non-small cell lung cancer (NSCLC);
* No history of malignancy within the past 5 years;
* Signed informed consent agreeing to participate in this study.

Exclusion Criteria:

* Unable to undergo surgical resection due to surgical contraindications;
* Postoperative pathology does not confirm non-small cell lung cancer (NSCLC), including but not limited to benign lesions, small cell lung cancer, metastatic tumors, or an insufficient or indeterminate histopathology report;
* History of malignancy within the past 5 years;
* Unable to obtain follow-up data;
* Refusal to sign the informed consent or withdrawal of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will retrospectively enroll 450 consecutive patients with stage IA~IIIB non-small cell lung cancer performed sleeve lobectomy in minimally invasive surgical techniques (RATS or VATS) from January 2015 to September 2024 in all three related centers. Baseline clinical information, surgery-related data, short-term postoperative outcomes, and long-term survival data (3-year OS and RFS) will be collected and analyzed using the propensity score matching method.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year RFS | 3 years
  In this study, the investigators will focus on the 3-year recurrence-free survival (RFS) of the participants between the two groups (RATS vs. VATS) for the comparison of the long-term oncologic outcomes, as the primary outcome.

SECONDARY OUTCOMES:
3-year OS | 3 years
  The investigators will also focus on the 3-year overall survival (OS) of the participants between the two groups (RATS vs. VATS) for the comparison of the long-term oncologic outcomes, as the secondary outcome.

OTHER OUTCOMES:
Intraoperative blood loss | up to 90 days
  The intraoperative blood loss will be investigated between RATS versus VATS sleeve lobectomy as one of the perioperative outcomes, measured in milliliter (mL).
Operative time | up to 90 days
  The operative time will be investigated between RATS versus VATS sleeve lobectomy as one of the perioperative outcomes, measured in minute (min).
Length of hospital stay | up to 90 days
  The length of hospital stay will be investigated between RATS versus VATS sleeve lobectomy as one of the perioperative outcomes, measured in day.
Postoperative drainage | up to 90 days
  The postoperative drainage will be investigated between RATS versus VATS sleeve lobectomy as one of the perioperative outcomes, measured in milliliter (mL).
Postoperative complications | up to 90 days
  The postoperative complications will be investigated between RATS versus VATS sleeve lobectomy as one of the perioperative outcomes, showed in the number of the participants who occurred postoperative complications (n).
Perioperative mortality | up to 90 days
  The perioperative mortality will be investigated between RATS versus VATS sleeve lobectomy as one of the perioperative outcomes, showed in the number of the participants who died within 90 days of surgery (n).
Number of dissected lymph nodes | up to 90 days
  The number of dissected lymph nodes will be investigated between RATS versus VATS sleeve lobectomy as one of the perioperative outcomes (n).
Margin status | up to 90 days
  The margin status will be investigated between RATS versus VATS sleeve lobectomy as one of the perioperative outcomes, showed in the number of the participants who had the positive or negative surgical margins (n).

CONTACTS AND LOCATIONS:
Overall Officials: Haifeng Shen, M.D., Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Xinghua Cheng, M.D. Ph.D., Study Director — Shanghai Chest Hospital of Shanghai Jiao Tong University; Yuhan Zhou, M.D., Study Director — Sir Run Run Shaw Hospital; Junqiang Fan, M.D., Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (3):
- China (3):
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Sir Run Run Shaw Hospital, Medical College, Zhejiang University, Hangzhou
  - Shanghai Chest Hospital, Shanghai Jiao Tong University, Shanghai

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Qiu T, Zhao Y, Xuan Y, Qin Y, Niu Z, Shen Y, Jiao W. Robotic sleeve lobectomy for centrally located non-small cell lung cancer: A propensity score-weighted comparison with thoracoscopic and open surgery. J Thorac Cardiovasc Surg. 2020 Sep;160(3):838-846.e2. doi: 10.1016/j.jtcvs.2019.10.158. Epub 2019 Nov 22. PMID 31924355
- [Background] Chen T, Zhao W, Ji C, Luo J, Wang Y, Liu Y, Weder W, Fang W. Minimally invasive sleeve lobectomy for centrally located lung cancer: A real-world study with propensity-score matching. Front Oncol. 2023 Feb 1;13:1099514. doi: 10.3389/fonc.2023.1099514. eCollection 2023. PMID 36816921
- [Background] Deng J, Jiang L, Li S, Zhang L, Zhong Y, Xie D, Chen C. The learning curve of video-assisted thoracoscopic sleeve lobectomy in a high-volume pulmonary center. JTCVS Tech. 2021 Jul 20;9:143-152. doi: 10.1016/j.xjtc.2021.07.006. eCollection 2021 Oct. PMID 34647085
- [Background] Pan X, Gu C, Yang J, Shi J. Robotic double-sleeve resection of lung cancer: technical aspects. Eur J Cardiothorac Surg. 2018 Jul 1;54(1):183-184. doi: 10.1093/ejcts/ezy070. PMID 29579169
- [Background] Jiao W, Zhao Y, Qiu T, Xuan Y, Sun X, Qin Y, Liu A, Sui T, Cui J. Robotic Bronchial Sleeve Lobectomy for Central Lung Tumors: Technique and Outcome. Ann Thorac Surg. 2019 Jul;108(1):211-218. doi: 10.1016/j.athoracsur.2019.02.028. Epub 2019 Mar 21. PMID 30904403
- [Background] Cerfolio RJ. Robotic sleeve lobectomy: technical details and early results. J Thorac Dis. 2016 Mar;8(Suppl 2):S223-6. doi: 10.3978/j.issn.2072-1439.2016.01.70. No abstract available. PMID 26981274
- [Background] Gonzalez-Rivas D, Fernandez R, Fieira E, Rellan L. Uniportal video-assisted thoracoscopic bronchial sleeve lobectomy: first report. J Thorac Cardiovasc Surg. 2013 Jun;145(6):1676-7. doi: 10.1016/j.jtcvs.2013.02.052. Epub 2013 Mar 15. No abstract available. PMID 23507125
- [Background] Shen H, Wang X, Nie Y, Zhang K, Wei Z, Yang F, Wang J, Chen K. Minimally invasive surgery versus thoracotomy for resectable stage II and III non-small-cell lung cancers: a systematic review and meta-analysis. Eur J Cardiothorac Surg. 2021 May 8;59(5):940-950. doi: 10.1093/ejcts/ezaa437. PMID 33370437
- [Background] Pages PB, Mordant P, Renaud S, Brouchet L, Thomas PA, Dahan M, Bernard A; Epithor Project (French Society of Thoracic and Cardiovascular Surgery). Sleeve lobectomy may provide better outcomes than pneumonectomy for non-small cell lung cancer. A decade in a nationwide study. J Thorac Cardiovasc Surg. 2017 Jan;153(1):184-195.e3. doi: 10.1016/j.jtcvs.2016.09.060. Epub 2016 Oct 13. PMID 27814899
- [Background] Ma Z, Dong A, Fan J, Cheng H. Does sleeve lobectomy concomitant with or without pulmonary artery reconstruction (double sleeve) have favorable results for non-small cell lung cancer compared with pneumonectomy? A meta-analysis. Eur J Cardiothorac Surg. 2007 Jul;32(1):20-8. doi: 10.1016/j.ejcts.2007.03.018. Epub 2007 Apr 17. PMID 17442581
- [Background] Riely GJ, Wood DE, Ettinger DS, Aisner DL, Akerley W, Bauman JR, Bharat A, Bruno DS, Chang JY, Chirieac LR, DeCamp M, Desai AP, Dilling TJ, Dowell J, Durm GA, Gettinger S, Grotz TE, Gubens MA, Juloori A, Lackner RP, Lanuti M, Lin J, Loo BW, Lovly CM, Maldonado F, Massarelli E, Morgensztern D, Mullikin TC, Ng T, Owen D, Owen DH, Patel SP, Patil T, Polanco PM, Riess J, Shapiro TA, Singh AP, Stevenson J, Tam A, Tanvetyanon T, Yanagawa J, Yang SC, Yau E, Gregory KM, Hang L. Non-Small Cell Lung Cancer, Version 4.2024, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2024 May;22(4):249-274. doi: 10.6004/jnccn.2204.0023. PMID 38754467
- [Background] Bender E. Epidemiology: The dominant malignancy. Nature. 2014 Sep 11;513(7517):S2-3. doi: 10.1038/513S2a. No abstract available. PMID 25208070
- [Background] Xia C, Dong X, Li H, Cao M, Sun D, He S, Yang F, Yan X, Zhang S, Li N, Chen W. Cancer statistics in China and United States, 2022: profiles, trends, and determinants. Chin Med J (Engl). 2022 Feb 9;135(5):584-590. doi: 10.1097/CM9.0000000000002108. PMID 35143424
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751